CLINICAL TRIAL: NCT02018302
Title: Post Study Continuation of C7 for G1D
Status: No longer available | Type: Expanded Access
Sponsor: Juan Pascual (Other)
Responsible Party: Sponsor-Investigator, Juan Pascual, Associate Professor, Director of the Rare Brain Disorders Program, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: UTSW 082013-016
Record Dates: First submitted 2013-12-11; First posted 2013-12-23 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Glut1 Deficiency Syndrome; Glucose Transporter Type 1 Deficiency Syndrome
Keywords: G1D; Glut1 Deficiency; Glucose Transporter Type 1 Deficiency; Glucose Transporter Type I Deficiency
MeSH Terms: conditions — Glut1 Deficiency Syndrome | interventions — triheptanoin

INTERVENTIONS:
Drug: Triheptanoin
  Other Names: C7 oil; Heptanoate; heptanoic acid

SUMMARY:
This protocol provides ongoing access to triheptanoin for patients who did complete an initial pilot protocol, and provides the opportunity to collect long-term safety data from patients treated with triheptanoin.

DETAILED DESCRIPTION:
Only patients who completed the initial pilot study were eligible. The study is ongoing with these patients only.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the pilot trial (UTSW 122010-186)

Exclusion Criteria:

* Subjects who did not complete the pilot trial (UTSW 122010-186)

Ages: 1 Month to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Pascual, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Marin-Valencia I, Good LB, Ma Q, Malloy CR, Pascual JM. Heptanoate as a neural fuel: energetic and neurotransmitter precursors in normal and glucose transporter I-deficient (G1D) brain. J Cereb Blood Flow Metab. 2013 Feb;33(2):175-82. doi: 10.1038/jcbfm.2012.151. Epub 2012 Oct 17. PMID 23072752
- [Background] Marin-Valencia I, Good LB, Ma Q, Duarte J, Bottiglieri T, Sinton CM, Heilig CW, Pascual JM. Glut1 deficiency (G1D): epilepsy and metabolic dysfunction in a mouse model of the most common human phenotype. Neurobiol Dis. 2012 Oct;48(1):92-101. doi: 10.1016/j.nbd.2012.04.011. Epub 2012 Apr 23. PMID 22683290
- [Background] Marin-Valencia I, Roe CR, Pascual JM. Pyruvate carboxylase deficiency: mechanisms, mimics and anaplerosis. Mol Genet Metab. 2010 Sep;101(1):9-17. doi: 10.1016/j.ymgme.2010.05.004. Epub 2010 Jun 9. PMID 20598931
- [Background] Wang D, Sands T, Tang M, Monani U, De Vivo D. Glucose Transporter Type 1 Deficiency Syndrome. 2002 Jul 30 [updated 2025 Mar 6]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1430/ PMID 20301603
- [Background] Perez-Duenas B, Prior C, Ma Q, Fernandez-Alvarez E, Setoain X, Artuch R, Pascual JM. Childhood chorea with cerebral hypotrophy: a treatable GLUT1 energy failure syndrome. Arch Neurol. 2009 Nov;66(11):1410-4. doi: 10.1001/archneurol.2009.236. PMID 19901175
- [Background] Jeffrey FM, Marin-Valencia I, Good LB, Shestov AA, Henry PG, Pascual JM, Malloy CR. Modeling of brain metabolism and pyruvate compartmentation using (13)C NMR in vivo: caution required. J Cereb Blood Flow Metab. 2013 Aug;33(8):1160-7. doi: 10.1038/jcbfm.2013.67. Epub 2013 May 8. PMID 23652627
- [Background] Xu F, Liu P, Pascual JM, Xiao G, Lu H. Effect of hypoxia and hyperoxia on cerebral blood flow, blood oxygenation, and oxidative metabolism. J Cereb Blood Flow Metab. 2012 Oct;32(10):1909-18. doi: 10.1038/jcbfm.2012.93. Epub 2012 Jun 27. PMID 22739621
- [Background] Pascual JM, Campistol J, Gil-Nagel A. Epilepsy in inherited metabolic disorders. Neurologist. 2008 Nov;14(6 Suppl 1):S2-S14. doi: 10.1097/01.nrl.0000340787.30542.41. PMID 19225367
- [Background] Wang D, Yang H, Shi L, Ma L, Fujii T, Engelstad K, Pascual JM, De Vivo DC. Functional studies of the T295M mutation causing Glut1 deficiency: glucose efflux preferentially affected by T295M. Pediatr Res. 2008 Nov;64(5):538-43. doi: 10.1203/PDR.0b013e318184d2b5. PMID 18614966
- [Background] Gomez Lado C, Couce Pico ML, Sanchez-Salmon A, Pascual JM. [Glucose transporter type 1 deficiency: a treatable neuro-metabolic disorder]. An Pediatr (Barc). 2008 Sep;69(3):285-6. doi: 10.1157/13125831. No abstract available. Spanish. PMID 18775281
- [Background] Pascual JM, Wang D, Yang R, Shi L, Yang H, De Vivo DC. Structural signatures and membrane helix 4 in GLUT1: inferences from human blood-brain glucose transport mutants. J Biol Chem. 2008 Jun 13;283(24):16732-42. doi: 10.1074/jbc.M801403200. Epub 2008 Apr 3. PMID 18387950
- [Background] Pascual JM, Wang D, Hinton V, Engelstad K, Saxena CM, Van Heertum RL, De Vivo DC. Brain glucose supply and the syndrome of infantile neuroglycopenia. Arch Neurol. 2007 Apr;64(4):507-13. doi: 10.1001/archneur.64.4.noc60165. Epub 2007 Feb 12. PMID 17296829
- [Background] Pascual JM. [Glucose transport hereditary diseases]. Med Clin (Barc). 2006 Nov 11;127(18):709-14. doi: 10.1157/13095099. Spanish. PMID 17169300
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Mao X, Cheng J, Yoo J, Noebels JL, De Vivo DC. A mouse model for Glut-1 haploinsufficiency. Hum Mol Genet. 2006 Apr 1;15(7):1169-79. doi: 10.1093/hmg/ddl032. Epub 2006 Feb 23. PMID 16497725
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Jhung S, Sun RP, De Vivo DC. Glut-1 deficiency syndrome: clinical, genetic, and therapeutic aspects. Ann Neurol. 2005 Jan;57(1):111-8. doi: 10.1002/ana.20331. PMID 15622525
- [Background] Pascual JM, Lecumberri B, Wang D, Yang R, Engelstad K, De Vivo DC. [Type 1 glucose transporter (Glut1) deficiency: manifestations of a hereditary neurological syndrome]. Rev Neurol. 2004 May 1-15;38(9):860-4. Spanish. PMID 15152356
- [Background] Pascual JM, Wang D, Lecumberri B, Yang H, Mao X, Yang R, De Vivo DC. GLUT1 deficiency and other glucose transporter diseases. Eur J Endocrinol. 2004 May;150(5):627-33. doi: 10.1530/eje.0.1500627. PMID 15132717
- [Background] Wang D, Pascual JM, Iserovich P, Yang H, Ma L, Kuang K, Zuniga FA, Sun RP, Swaroop KM, Fischbarg J, De Vivo DC. Functional studies of threonine 310 mutations in Glut1: T310I is pathogenic, causing Glut1 deficiency. J Biol Chem. 2003 Dec 5;278(49):49015-21. doi: 10.1074/jbc.M308765200. Epub 2003 Sep 16. PMID 13129919
- [Background] Pascual JM, Van Heertum RL, Wang D, Engelstad K, De Vivo DC. Imaging the metabolic footprint of Glut1 deficiency on the brain. Ann Neurol. 2002 Oct;52(4):458-64. doi: 10.1002/ana.10311. PMID 12325075
- [Background] Iserovich P, Wang D, Ma L, Yang H, Zuniga FA, Pascual JM, Kuang K, De Vivo DC, Fischbarg J. Changes in glucose transport and water permeability resulting from the T310I pathogenic mutation in Glut1 are consistent with two transport channels per monomer. J Biol Chem. 2002 Aug 23;277(34):30991-7. doi: 10.1074/jbc.M202763200. Epub 2002 May 24. PMID 12032147
- [Background] De Vivo DC, Wang D, Pascual JM, Ho YY. Glucose transporter protein syndromes. Int Rev Neurobiol. 2002;51:259-88. doi: 10.1016/s0074-7742(02)51008-4. No abstract available. PMID 12420362
- [Background] Brockmann K, Wang D, Korenke CG, von Moers A, Ho YY, Pascual JM, Kuang K, Yang H, Ma L, Kranz-Eble P, Fischbarg J, Hanefeld F, De Vivo DC. Autosomal dominant glut-1 deficiency syndrome and familial epilepsy. Ann Neurol. 2001 Oct;50(4):476-85. doi: 10.1002/ana.1222. PMID 11603379